CLINICAL TRIAL: NCT05874037
Title: Fluvoxamine as a Treatment for Long COVID-19: A Randomized Placebo Controlled Trial
Brief Title: Fluvoxamine for Long COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Balvi COVID Fund (Unknown); BJH Townley Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202211024
Record Dates: First submitted 2023-05-22; First posted 2023-05-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluvoxamine (Experimental)
  Interventions: Drug: Fluvoxamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Fluvoxamine

INTERVENTIONS:
Drug: Fluvoxamine — Fluvoxamine is an FDA approved drug for the treatment of OCD. This trial is testing the effects of the drug on long COVID.

SUMMARY:
This clinical trial aims to test the effects of fluvoxamine as a treatment for Long COVID. Fluvoxamine is an FDA approved SSRI for Obsessive Compulsive Disorder (OCD), that has already had success in preventing hospitalization in patients with COVID-19 (STOP COVID and TOGETHER trials). This trial is testing whether fluoxamine helps to improve symptoms and the negative impacts of long COVID in residents of Missouri and Illinois.

DETAILED DESCRIPTION:
This clinical trial will test a promising drug for treatment of long COVID in 300 adults who 1) are post-COVID-19 (at least 3 months since initial COVID symptoms and/or test confirming SARS-CoV-2 infection); and 2) have evidence of neurocognitive Long COVID (e.g., "brain fog", trouble concentrating, etc) which is causing suffering and/or impairment. The trial will determine whether fluvoxamine (1) reduces long COVID symptoms, 2) improves cognitive performance. Fluvoxamine is an SSRI (FDA approved for OCD) that also activates the sigma-1 receptor (an immunomodulatory receptor). It has been shown to prevent clinical deterioration and hospitalization in outpatients with acute COVID-19 (STOP COVID and TOGETHER trials). For the current study, we will randomize participants to fluvoxamine which is initially dosed at their preference, vs. placebo. This is done in the following manner. First, each participant will receive an acute bout of fluvoxamine: one dose of 25mg, then one dose of 50mg, then one dose of 100mg. We will assess their subjective reaction to these test doses and use the information to randomize them to an individually tailored course of fluvoxamine, vs. a matched placebo, for 16 weeks. The benefits of this are (1) participants are more likely to accept randomization and continue in the study if randomized to a dose they've already tested and accepted; (2) participants' initial response, if any, to the acute dose may allow future precision-medicine use of fluvoxamine, allowing physicians to give patients a test dose and then a full trial preferentially to participants who are likely to respond. After the randomized portion of the trial, participants will be given an opportunity to participate in open-label treatment with fluvoxamine for 16 weeks. At the end of treatment, the study medication will be tapered off over an approximate 1-2 week period, depending on the final dose of study medication, and adjusted as appropriate if they experience discontinuation symptoms. Outcome assessments will be a combination of patient-reported assessments and validated neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

1. Men and woman age 25 and older;
2. Not currently hospitalized
3. Participant self-report of past acute COVID episode with symptom onset and/or initial positive test at least 3 months since initial COVID symptoms and/or test confirming SARS-CoV-2 infection Note: Since some people with long COVID may not have been able to obtain testing during the acute phase of illness, history of a positive COVID-19 test is not required. We will collect data regarding the results of any past COVID-19 testing, but this will not affect eligibility for the trial.
4. Currently symptomatic with self-reported worsening of cognitive function for at least the past 2 months, that could not be better explained by other reasons (i.e. alternative diagnosis or medication changes).
5. Able to provide informed consent.
6. Currently reside in Missouri or Illinois

Exclusion Criteria:

1. Illness severe enough to require hospitalization at the time of starting the study.
2. Unstable medical comorbidities (eg decompensated cirrhosis), per patient report and/or medical records.
3. Immunocompromised from the following: solid organ transplant, BMT, high dose steroids (>20mg prednisone per day), or tocilizumab
4. Already enrolled in another COVID 19 medication trial (not including vaccination or prophylaxis trials)
5. Unable to provide informed consent
6. Unable to perform the study procedures, including not being a resident of the states of Missouri or Illinois
7. Taking donepezil (rationale: donepezil is a S1R agonist), or sertraline (rationale: sertraline is a strong sigma-1 antagonist).
8. Taking phenytoin (rationale: fluvoxamine inhibits its metabolism), clopidogrel (rationale: fluvoxamine inhibits its metabolism from pro-drug to active drug which raises risk of cardiovascular events), and St John's wort (rationale: fluvoxamine + St John's wort are considered contraindicated because of the risk of serotonin syndrome)
9. Taking SSRIs or SNRIs.
10. Individuals who report they have bipolar disorder or are taking medication for bipolar disorder (lithium, valproate, high-dose antipsychotic), unless the investigator concludes that the risk for mania is unlikely (ie it is doubtful that the patient actually has bipolar disorder).
11. Individuals who take alprazolam or diazepam and are unwilling to cut the medication by 25% (rationale: fluvoxamine modestly inhibits the metabolism of these drugs).
12. Participants taking theophylline, tizanidine, clozapine, or olanzapine (drugs with a narrow therapeutic index that are primarily metabolized by CYP 1A2, which is inhibited by fluvoxamine) will be reviewed with a study investigator and excluded unless the investigator concludes that the risk to the participant is low (this would be unlikely; example: participant takes tizanidine only as needed and is willing to avoid it during study duration).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Total of symptom score via the daily questionnaire | Approximately 18 weeks
  Improvement in combined total score based upon the self-report daily questionnaire which asks about trouble concentrating, anxiety, depression and fatigue. Respondents rate how much of a problem the symptom is "right now" on a scale of 0 (no problem) to 100 (severe problem).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided